CLINICAL TRIAL: NCT01177605
Title: Assessment of Efficacy and Tolerance of a Follow-On Milk Containing a Mixture of Prebiotics Fed to Young Children in Salvador, Bahia, Brazil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Other Study IDs: 3376-1 (8575)
Record Dates: First submitted 2010-08-03; First posted 2010-08-09 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Gastrointestinal Problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vanilla flavored milk-based beverage containing no prebiotics (Placebo Comparator): Vanilla flavored milk-based beverage containing no prebiotics
  Interventions: Other: Nutritional vanilla flavored beverage - 1) Milk-based beverage containing prebiotics 2) Milk-based beverage containing no prebiotics
- Vanilla flavored milk-based beverage containing prebiotics (Experimental): Vanilla flavored milk-based beverage containing prebiotics
  Interventions: Other: Nutritional vanilla flavored beverage - 1) Milk-based beverage containing prebiotics 2) Milk-based beverage containing no prebiotics

INTERVENTIONS:
Other: Nutritional vanilla flavored beverage - 1) Milk-based beverage containing prebiotics 2) Milk-based beverage containing no prebiotics — Nutritional vanilla flavored beverage - 1) Milk-based beverage containing prebiotics 2) Milk-based beverage containing no prebiotics

SUMMARY:
This clinical study will evaluate the effect on incidence of diarrhea, respiratory illness, stool patterns and growth of two cow's milk-based beverages for children.

ELIGIBILITY:
Inclusion Criteria:

* Child 9 - 48 months of age
* Child has consumed a cow follow-on milk during the 48 hours prior to enrollment
* Child's weight for age is within the 10th -90th percentiles
* Child's length for age is within 10th - 90th percentiles
* Signed informed consent obtained

Exclusion Criteria:

* Children who are receiving predominantly breast-milk
* Serious concurrent illness
* Children with diarrhea or acute respiratory infection during the 48 hours prior to randomization
* Children with a history of underlying metabolic or chronic disease or congenital malformation which, in the opinion of the Investigator, is likely to interfere with the normal growth and development or the evaluation of the participant.

Ages: 9 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 2006-09; Primary Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Bahia School of Medicine, Salvador, Estado de Bahia, Brazil